CLINICAL TRIAL: NCT05424159
Title: Prospective Phase II Clinical Trial of Ablative Carbon Ion Radiotherapy With Pencil Beam Scanning Using Simultaneous Integrated Boost for Locally Advanced Unresectable Pancreatic Cancer
Brief Title: Ablative Carbon Ion Radiotherapy With Pencil Beam Scanning for Locally Advanced Unresectable Pancreatic Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Proton and Heavy Ion Center (Other)
Responsible Party: Principal Investigator, Guoliang Jiang, Principal Investigator, Shanghai Proton and Heavy Ion Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPHIC-TR-PaCa2022-01
Record Dates: First submitted 2022-06-10; First posted 2022-06-21 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-06

CONDITIONS: Pancreatic Cancer Non-resectable
Keywords: Locally advanced unresectable pancreatic cancer; Carbon ion radiotherapy; Phase II clinical trial; Ablative dose; Optimized linear energy transfer
MeSH Terms: interventions — Heavy Ion Radiotherapy

STUDY DESIGN:
Intervention Model Description: Radiation: carbon ion radiotherapy for tumors without invasion of GI
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with locally advanced unresectable pancreatic cancer (Experimental): Patients with locally advanced unresectable pancreatic cancer without invasion of the gastrointestinal tract, cT4N0-2M0 Stage III (AJCC/UICC Version 8).
  Interventions: Radiation: Carbon ion radiotherapy

INTERVENTIONS:
Radiation: Carbon ion radiotherapy — Patients with locally advanced unresectable pancreatic cancer without invasion of gastrointestinal tract will received ablative carbon ion radiotherapy. The prescription dose for primary pancreatic lesion, positive lymph node, and retroperitoneal high-risk recurrence area is 67.5 Gy (RBE weighted dose) in 15 fractions for 3 weeks; Pancreatic primary lesion and positive lymph node SIB to 75 Gy (RBE weighted dose) in 15 fractions for 3 weeks.

SUMMARY:
The aim of this study is to investigate the clinical efficacy and safety of ablative carbon ion radiotherapy for locally advanced unresectable pancreatic cancer with pencil beam scanning and simultaneous integrated boost (SIB) technology.

DETAILED DESCRIPTION:
The aim of this study is to investigate the clinical efficacy and safety of ablative carbon ion radiotherapy for locally advanced unresectable pancreatic cancer using pencil beam scanning and simultaneous integrated boost technology with respect to toxicity and tumor control. All enrolled patients will receive carbon ion radiotherapy for the primary pancreatic lesions, positive lymph nodes, and retroperitoneal high-risk recurrence areas. The prescription dose for primary pancreatic lesion, positive lymph node, and retroperitoneal high-risk recurrence area is 67.5 Gy (RBE weighted dose) in 15 fractions for 3 weeks; Pancreatic primary lesion and positive lymph node SIB to 75 Gy (RBE weighted dose) in 15 fractions for 3 weeks. The primary endpoint is 2-year cumulative local regional progression rate (LRP), and the secondary endpoint is to assess the overall survival (OS) and toxicities. Toxicity was assessed using the Common Adverse Event Evaluation Criteria (CTCAE) Version 5.0, and safety and toxicity will be assessed by clinical examination, laboratory examination, and imaging (including CT, MRI, and/or PET/CT).

ELIGIBILITY:
Inclusion Criteria:

1. Have the ability to sign the written informed consent;
2. Ductal adenocarcinoma of the pancreas confirmed by histopathology or cytopathology;
3. Distant metastasis was excluded by imaging assessment (PET-CT, cranial MRI), and was defined as locally advanced unresectable according to NCCN Guidelines Version 2022.1, that is, T4N0-2M0, Stage III (AJCC/UICC Version 8);
4. The maximum diameter of pancreatic primary lesion and positive lymph node ≤7cm;
5. Pancreas primary lesion or positive lymph node did not invade digestive tract (stomach, duodenum and small intestine);
6. Eastern Cooperative Oncology Group (ECOG) performance score 0-1;
7. Adequate bone marrow function (neutrophil count ≥1.5×109/L, platelet count ≥100×109/L, hemoglobin ≥10.0g/dL);
8. Adequate liver function (total bilirubin <1.5 times the upper limit of normal value, aminotransferase <2.5 times the upper limit of normal value);
9. Adequate renal function (serum creatinine <2mg/dL, or creatinine clearance >50mL/min).

Exclusion Criteria:

1. Multiple primary pancreatic lesions (>1);
2. Tumor invaded the adjacent digestive tract;
3. Radiation therapy history;
4. Other local treatments history for pancreatic cancer, such as HIFU and irreversible electroporation;
5. The irradiation dose of organs at risk cannot reach the dose constraint;
6. Other malignant tumors history;
7. Inability to understand the purpose of treatment or unwillingness/inability to sign informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
2-year cumulative local regional progression rate (LRP) | From the date of the initiation of radiotherapy until the date of first documented occurrence of local regional progression, assessed up to 24 months.
  LRP was defined as the percentage of patients with local disease progression (within irradiated area) in the intentional population.

SECONDARY OUTCOMES:
2-year Overall survival (OS) | From the date of diagnosis until the date of death from any cause, assessed up to 24 months.
  OS was defined as the percentage of patients dead in the intentional population.
Acute toxicity | From the date of the initiation of radiotherapy until the date of 3 months after radiotherapy.
  Toxicity was assessed using Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. Safety and toxicity will be assessed by clinical examination, laboratory examination, and imaging (including CT, MRI, and/or PET/CT).
Late toxicity | 3 months after radiotherapy.
  Toxicity was assessed using Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. Safety and toxicity will be assessed by clinical examination, laboratory examination, and imaging (including CT, MRI, and/or PET/CT).

CONTACTS AND LOCATIONS:
Overall Officials: Zheng Wang, MD, PhD, Principal Investigator — Shanghai Proton and Heavy Ion Center; Xin Cai, MD, Principal Investigator — Shanghai Proton and Heavy Ion Center
Locations (1):
- Shanghai Proton and Heavy Ion Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: No